CLINICAL TRIAL: NCT02006303
Title: Prostatic Artery Embolization Versus 532 nm Green Light Laser Photoselective Vaporization of the Prostate for Treating Catheter-Dependent Patients With Benign Prostatic Hyperplasia: A Randomized Controlled Clinical Study
Brief Title: Prostatic Artery Embolization Versus 532 nm Green Light PVP for Catheterized Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Victoria Hospital, Canada (Other)
Responsible Party: Principal Investigator, Mostafa Elhilali, Professor of Urology, Royal Victoria Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-100-SDR
Record Dates: First submitted 2013-11-28; First posted 2013-12-10 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Benign Prostate Hyperplasia; Urinary Retention
Keywords: Benign Prostate Hyperplasia; Green light; Photoselective vaporization of the prostate; Prostatic artery embolization; Outcome
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Retention | interventions — Photoelectron Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Green light PVP (Active Comparator): The KTP:YAG laser is based on the principle of passing Nd:YAG laser light through a KTP crystal. This halves the wavelength of the emitted laser to 532 nm and doubles its frequency. The emitted light is a visible green light, which is strongly absorbed by red tissues and hemoglobin; this renders a blood rich organ such as the prostate gland to be an excellent target. Prostate tissue is vaporized leaving an appropriate cavity for voiding.
  Interventions: Procedure: Green light PVP
- Prostatic Artery Embolization (Active Comparator): Prostatic artery embolization consists of gaining access into the patients arterial system via a common femoral artery puncture using a small needle and sheath. Once the access is established, a micro-catheter is navigated through the arterial system using X-ray guidance into the arteries feeding the prostate. There, small polyvynil alcohol plastic beads are injected to block the blood flow to the prostate. By doing so, the prostate undergoes an ischemic injury and there is reduction in gland size and relief of obstructive symtpoms.
  Interventions: Procedure: Prostatic artery embolization

INTERVENTIONS:
Procedure: Green light PVP — The green light laser has a wavelength of 532 nm which is strongly absorbed by red tissues and hemoglobin; this renders a blood rich organ such as the prostate gland to be an excellent target. The procedure uses the technology of high-powered laser light combined with fiber optics to vaporize the overgrowth of prostate cells quickly and accurately. As the surgeon directs the laser at the prostate, the intense pulses of light emitted from the fiber are absorbed by the blood. Within moments, the temperature of the blood becomes so great it causes the nearby cells to vaporize. Once the procedure is completed, patients have immediate post-operative symptom relief and dramatic improvements in symptoms, urinary flow rates, and bladder emptying.
  Other Names: XPS (Xcelerated Performance System); PVP; Photoselective vaporization of the prostate
  Arms: Green light PVP
Procedure: Prostatic artery embolization — Prostatic artery embolization consists of gaining access into the patients arterial system via a common femoral artery puncture using a small needle and sheath. Once the access is established, a micro-catheter is navigated through the arterial system using X-ray guidance into the arteries feeding the prostate. There, small polyvynil alcohol plastic beads are injected to block the blood flow to the prostate. By doing so, the prostate undergoes an ischemic injury and there is reduction in gland size and relief of obstructive symtpoms.
  Other Names: PAE
  Arms: Prostatic Artery Embolization

SUMMARY:
The primary objective is to assess whether prostatic artery embolization has a similar efficacy and safety profile as GreenLight PVP in treating patients with urinary retention secondary to benign prostate hyperplasia (BPH). Subjects who consent will be randomized to either the Prostate embolization (PAE) arm or to the GreenLight PVP arm.

The primary endpoint of efficacy of the procedure is measured by the ability of the patient to void. The secondary endpoints recorded will include patients' satisfaction measured by International Prostate Symptom Score (IPSS), peak flow rate (Qmax) and post-void residual urine volume (PVR) and prostate specific antigen (PSA) will be measured at 3, 6, and 12 months post treatment. Also, reduction in prostate volume is considered by MRI preoperatively, 3 months and 12 months.

DETAILED DESCRIPTION:
The primary objective is to assess whether prostatic artery embolization has a similar efficacy and safety profile compared to GreenLight PVP in treating patients with urinary retention secondary to benign prostate hyperplasia (BPH) that have failed medical management.

The target population is composed of subjects referred to the urology department for treatment of BPH who have failed medical treatment, who present with permanent bladder catheterization and who meet the eligibility criteria.

Subjects who consent will be randomized to either the Prostate embolization (PAE) arm or to the GreenLight PVP arm.

The primary endpoint of efficacy of the procedure is measured by the successful removal of bladder catheter and ability of the patient to void. As well, the secondary endpoints recorded will be: International Prostate Symptom Score (IPSS), peak flow rate (Qmax) and post-void residual urine volume (PVP) and prostate specific antigen (PSA) will be measured at 3, 6, and 12 months post treatment. Trans-rectal ultrasound (TRUS) will be performed for measurement of prostate volume for the stratified randomization process. All adverse events will be captured and analyzed. MRI will be performed preoperatively, 3 months and 12 months. Hospital stays after the procedures will not be considered serious adverse events, unless a hospital admission occurs because of a complication of the treatment performed.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects, over 50 years of age at the time of enrollment.
2. Subjects referred to urology for BPH leading to permanent indwelling bladder catheters and are considered poor surgical candidates
3. Written informed consent to participate in the study.
4. Ability to comply with the requirements of the study procedures

Exclusion Criteria:

1. Previous surgical treatment for BPH
2. Presence of bladder stones
3. History of prostate cancer
4. Prostate size > 150 g
5. History of urethral stenosis or its management
6. Known of suspected neurogenic bladder
7. History of recent hematochezia in the last 3 months
8. Contraindication to intravascular iodinated contrast such as allergies or significant elevated creatinine/renal failure
9. Uncorrected coagulopathy
10. Subjects who participated in an active stage of any drug, intervention or treatment trial within 30 days of enrollment.
11. Subjects with preexisting conditions, which, in the opinion of the investigator, interfere with the conduct of the study.
12. Subjects who are uncooperative or cannot follow instructions.
13. Mental state that may preclude completion of the study procedure or obtention of informed consent

Ages: 40 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Ability of the patient to void after removal of the urethral catheter | At 24-hours for PVP green light laser and 1-3 weeks for embolization

SECONDARY OUTCOMES:
Patient subjective satisfaction of both procedures evaluated by the International Prostate Symptom Score (IPSS) | At 3, 6, and 12 months post treatment
Degree of prostatic size reduction evaluated by MRI | Preoperatively, 3 months and 12 months.
Change in peak flow rate (Qmax) and | At 3, 6 and 12 months post treatment
Change in post-void residual urine volume (PVR) | At 3, 6, and 12 months
Change in prostate specific antigen (PSA) | At 3, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Elhilali, MD,PhD,FRCSC, Study Chair — Royal Victoria Hospital, Canada
Locations (2):
- Canada (2):
  - Royal Victoria Hospital, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec